CLINICAL TRIAL: NCT06330753
Title: Synergy Between Patient and Clinician: Using a Trauma-Informed Care Plan
Acronym: TICP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Annie Lewis-Oconnor, NP, Director of Research and Innovation, Center for Nursing Excellence, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000682
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Trauma and Stressor Related Disorders; Violence, Structural; Violence, Domestic; Violence, Sexual
Keywords: trauma; violence; abuse
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Coitus; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective study designed to explore the acceptability, intervention appropriateness of trauma-informed care plans and the feasibility of trauma-informed care plans by patients and members of the health care team
Masking Description: Participants (patients and providers) will be de-identified
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and Acceptability of Trauma-informed Care Plans (TICP) (Other): Per our IRB protocol - Patient participants and clinician participants will be asked (via a survey) to rate their:
  Acceptability of the Trauma-informed Care Plan, the Appropriateness of the TICP and the feasibility of the TICP. The intervention is the TICP place in the Electronic Medical Record right below the patient's name (on the Storyboard).
  Interventions: Other: Trauma-informed Care Plan-

INTERVENTIONS:
Other: Trauma-informed Care Plan- — Per our IRB protocol patient participates will be consented for this study. A member of the healthcare team ( licensed nurse, social worker or doctor) will conduct the TICP with the patient. The TICP will be placed in the electronic medical record right below the patients name. The workflow is such is that if any plan of care placed on the Storyboard (under the patient's name) should be read first before engaging with a patient.

SUMMARY:
The goal of this prospective study is to test the: acceptability of trauma-informed care plans; the intervention appropriateness; and the feasibility of the trauma-informed care plans in the electronic health care record. Patient seen in various health care settings and how have complex health care needs will be invited to participate in this study. The aims to are:

Aim 1: Explore the acceptability of trauma-informed care plans, the appropriateness of trauma-informed care plans, and the feasibility of Trauma-Informed Care Plans(TICP) when used by clinicians on the health care team (HCTC). Hypothesis 1: HCTC using the TICP will report its acceptability, feasibility, satisfaction and ease of use. Hypothesis 2: HCTC will report heightened awareness of intersection of trauma and social determinants of health. Hypothesis 3: HCTC will report more awareness of the patient's unique preferences and will be better informed regarding the unique plan of care for their patient.

Aim 2: Explore the impact of having a TICP by patients understanding how the TICP may have improved their experience around care and treatment. Hypothesis 1: patients will report: improved satisfaction with their care. Hypothesis 2: patients will report feeling better known by HCT. Hypothesis 3: will report less stress and anxiety related to health care encounters.

ELIGIBILITY:
Inclusion Criteria:

* patients ( ages 18-60)
* who have frequent health care appointments
* have complex health care needs
* consent to participate in study
* English or spanish speaking.

Exclusion Criteria:

* patients less than 18 and older than 60.
* patients too ill (medically/phytologically) to consent.
* suicidal or homicidal patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Trauma Informed Care Plans | 6-10 months
  This study is exploring the acceptability of trauma-informed care plans by the percentage of patients and clinicians that find the TICP acceptable

SECONDARY OUTCOMES:
Intervention Appropriateness of Trauma-Informed Care plans | 6-10 months
  This study is exploring the appropriateness of trauma-informed care plans by the percentage of patients and clinicians that find the TICP to be appropriate
Feasibility of the trauma-informed care plans | 6- 10 months
  This study is exploring the feasibility of the trauma-informed care plans by the percentage of patients and clinicians that find the trauma-informed care plans to be feasible.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States